CLINICAL TRIAL: NCT05814042
Title: Next Generation ORS: Randomized Controlled Trial Comparing ORS With Calcium vs Standard ORS in Reducing Severity With Acute Watery Diarrhea in Adults
Brief Title: Next Generation ORS: Controlled Trial Comparing ORS With Calcium vs Standard ORS in Reducing Severity of Acute Watery Diarrhea
Acronym: ORS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202202746 -N -R; 1R21AI169282-01A1 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-07

CONDITIONS: Diarrhea; Cholera
MeSH Terms: conditions — Diarrhea; Cholera | interventions — World Health Organization oral rehydration solution; Calcium

STUDY DESIGN:
Intervention Model Description: Two groups: Control vs Intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrient based intervention (Experimental): Nutrition supplement used to stop diarrhea
  Interventions: Drug: Next Generation ORS (oral rehydration solution) (including placebo
- Standard of Care oral rehydration solution (Active Comparator): Standard of care nutrition supplement used to stop diarrhea.
  Interventions: Drug: Current standard control ORS (oral rehydration solution)

INTERVENTIONS:
Drug: Next Generation ORS (oral rehydration solution) (including placebo — Nutrition used to stop diarrhea
  Other Names: WHO Reduced Osmolarity ORS with Calcium
  Arms: Nutrient based intervention
Drug: Current standard control ORS (oral rehydration solution) — current standard control ORS in diarrheic patients with cholera
  Other Names: WHO Reduced Osmolarity ORS
  Arms: Standard of Care oral rehydration solution

SUMMARY:
Diarrhea remains a leading killer of children in need of better treatments.

DETAILED DESCRIPTION:
Diarrhea remains a leading killer of children in need of better treatments. Oral Rehydration Solution (ORS) is currently the only oral therapy that is recommended for children with acute diarrhea. Although it is valuable for correcting dehydration and is considered the primary reason for the substantial reduction in mortality from diarrhea in children, ORS does not have the capacity to "halt" intestinal fluid loss and thus, does not offer a rapid relief of a child's diarrhea symptom, and its use by caregivers and medical practitioners has markedly dropped (estimate use in 1/3 of cases who need it). In recognition of its limitations, continuous efforts have been made to modify the composition of ORS. However, none has targeted the central diarrhea-causing pathways and produced a satisfactory outcome in children. New therapeutic approaches and methods are needed. The proposed new ORS is based on recent discovery of the first inclusive antidiarrheal mechanism in the intestine, CaSR (calcium-sensing receptor) that targets all known diarrhea causing pathways. It works in animals. This R21 is the 1st proof-of-concept clinical study in humans and is intended to investigate its safety and efficacy. Two Specific Aims are proposed to determine new ORS safety and efficacy in patients with diarrhea. In the safety study, the investigators propose to enroll 396 diarrheal adults (198 in Intervention New ORS group and 198 in standard WHO ORS). In the efficacy study, the investigators plan to enroll 396 diarrheal adults (198 in Intervention New ORS group and 198 in standard WHO ORS, these will be same patients employed for the safety study). These diarrheal patients will be recruited from the Dhaka area in Bangladesh. At the conclusion of the study, we expect to develop a novel oral rehydrating solution that is inexpensive and practical to use in all the countries. Hypothesis: the volume output Intervention should reduce stool weight/output of diarrhea by 30%.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, age between 18 and 60 years, history of acute watery diarrhea (defined as the passage of ≥3 loose or watery stools in the past 24 hours) for less than 24 h before admission, either signs of severe dehydration and stool positive for Vibrio cholerae, and successful rehydration with intravenous fluids within the first 6 h after admission (cholera group), or signs of some dehydration and stool negative for V. cholera (non-cholera group) , and successful rehydration with intravenous or oral fluids within the first 6 h

Exclusion Criteria:

* Pregnancy as determined by history of last menstrual period, bloody diarrhea, signs of systemic infection that needed intravenous antibiotics, or inability to rehydrate with intravenous fluid therapy in the first 6 h after admission.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stool Volume Output | Year 2
  Stool output is defined as the weight of stool in g per kg bodyweight after initial intravenous and or oral hydration

SECONDARY OUTCOMES:
Duration of diarrhea | year 2
  Duration of diarrhea is the time (in hour) from randomization until cessation of diarrhea
Stool frequency | year 2
  stool frequency is defined as the number of stool per day
Percentage of patients who vomit | year 2
  Percentage of patients who vomit from randomization until cessation of diarrhea
Percentage of patients who require unscheduled intravenous therapy | year 2
  Percentage of patients who require unscheduled intravenous therapy from randomization until cessation of diarrhea
Intake of ORS | year 2
  Intake of ORS (ml) from randomization until cessation of diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Sam Cheng, MD. PhD, Principal Investigator — University of Florida
Locations (1):
- ICDDR,B Dhaka Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT05814042/ICF_000.pdf